CLINICAL TRIAL: NCT04239300
Title: Efficiency and Safety of Water Birth in Maternity Hospitals in Uncomplicated Pregnancy.
Brief Title: Efficiency and Safety of Water Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akusherstvo Pro (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AlusherstvoPro
Record Dates: First submitted 2020-01-09; First posted 2020-01-27 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2020-03

CONDITIONS: Water Birth
Keywords: water birth
MeSH Terms: interventions — Parturition; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main group (Experimental): The participant in main group have water labour
  Interventions: Behavioral: Delivery in water
- Control group (No Intervention): The participant in control group will not have water labour

INTERVENTIONS:
Behavioral: Delivery in water — Participants delivery in water
  Arms: Main group

SUMMARY:
Water birth are not risks factors for newborns.

DETAILED DESCRIPTION:
Investigators will study medical records of woman who have water birth and evaluate different parameters. Study lasts from February 2020 till April 2021. The questionnaire contain information about woman's expectations of labour Number of participant is approximately 500.

ELIGIBILITY:
Inclusion Criteria:

* delivery alive newborn in water
* age 18-45
* single pregnancy

Exclusion Criteria:

* antenatal death
* dead fetus
* age under 18 and up 45
* multiple pregnancy
* somatic diseases
* preeclampsia
* mental diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1080 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Perineal trauma | 1 day
  The number and percentage of perineal trauma during labour

SECONDARY OUTCOMES:
Episiotomy | 1 day
  The number and percentage of episiotomy trauma during labour
Newborns wellbeing | 1 day
  Apgar scale
Infections complications from newborns | 3 days
  The number of Infections complications

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - OOO MD proect 2010, Ufa, Bashkortostan Republic
  - Schelkovo Perinatal Center, Moscow, Moscow Oblast

IPD SHARING:
Plan to Share IPD: Undecided